CLINICAL TRIAL: NCT00500760
Title: A Phase 2, Randomized Trial of Chemoradiation With or Without Panitumumab in Subjects With Unresected, Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Addition of Panitumumab to Chemoradiation Therapy in Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20062080
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; panitumumab
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Cisplatin; Panitumumab

ARMS (2):
- Panitumumab Plus Chemoradiation (Experimental): Participants received standard radiation therapy for 7 weeks and cisplatin 75 mg/m^2 and panitumumab 9 mg/kg on Days 1, 22 and 43.
  Interventions: Drug: Cisplatin; Radiation: Standard Fractionation Radiotherapy; Drug: Panitumumab
- Chemoradiotherapy Alone (Active Comparator): Participants received standard radiation therapy for 7 weeks and cisplatin 100 mg/m^2 on Days 1, 22, and 43.
  Interventions: Drug: Cisplatin; Radiation: Standard Fractionation Radiotherapy

INTERVENTIONS:
Drug: Cisplatin — Administered intravenously (IV; in a vein)
Radiation: Standard Fractionation Radiotherapy — 70 Gy administered in 2 Gy fractions daily for 5 days a week for 7 weeks (35 fractions)
Drug: Panitumumab — Administered intravenously
  Other Names: Vectibix®
  Arms: Panitumumab Plus Chemoradiation

SUMMARY:
The addition of chemotherapy to radiotherapy (chemoradiation) has improved outcomes for patients with locally advanced squamous cell carcinoma of the head and neck but additional improvements to treatment regimens are needed. The study is investigating if the addition of a targeted therapy (panitumumab) can improve the efficacy of chemoradiation without adding unmanageable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Stage III or IVa-b (M0) squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (you must be well enough to receive chemoradiation therapy)
* You must be at least 18 years of age
* Your test results must show that your kidneys, liver and blood cells are working adequately and that, if you are female, you are not pregnant
* You must have measurable disease

Exclusion Criteria:

* Cancer of the nasopharynx, sinus, salivary gland or skin
* History of another cancer (other than head and neck) unless treated with curative intent and with no evidence of disease for more than 3 years, with the exception of non-melanoma skin cancer or in situ cervical cancer
* Previous treatment with anti-endothelial growth factor receptor (EGFr) antibody therapy or EGFr inhibitors
* Previous treatment for head and neck cancer, with chemotherapy, surgery (except nodal sampling or biopsy) or radiotherapy
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within one year before you join the study
* Chronic obstructive pulmonary disease (pneumonia or respiratory decompensation) resulting in hospitalization within 6 months of study screening
* History or evidence of interstitial lung disease (e.g. pneumonitis or pulmonary fibrosis)
* Major surgery within 28 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2011-03-29 (Actual); Study Completion 2011-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Mesia R, Henke M, Fortin A, Minn H, Yunes Ancona AC, Cmelak A, Markowitz AB, Hotte SJ, Singh S, Chan AT, Merlano MC, Skladowski K, Zhang A, Oliner KS, VanderWalde A, Giralt J. Chemoradiotherapy with or without panitumumab in patients with unresected, locally advanced squamous-cell carcinoma of the head and neck (CONCERT-1): a randomised, controlled, open-label phase 2 trial. Lancet Oncol. 2015 Feb;16(2):208-20. doi: 10.1016/S1470-2045(14)71198-2. Epub 2015 Jan 15. PMID 25596660
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 153 patients were enrolled with 89 patients on panitumumab plus chemoradiation arm, and 64 patients on chemoradiotherapy alone arm.
Groups:
- Panitumumab Plus Chemoradiation: Participants received standard radiation therapy for 7 weeks, cisplatin 75 mg/m^2 and panitumumab 9 mg/kg intravenously on Days 1, 22 and 43.
Period: Overall Study
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Started | 89 | 64
Received Treatment | 87 | 63
Completed | 46 | 40
Not Completed | 43 | 24
Not completed — Death | 32 | 15
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Administrative decision | 2 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone | Total
Number analyzed (Participants) | 89 | 64 | 153
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (8.4) | 56.6 (8.8) | 57.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 76 | 57 | 133
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 82 | 55 | 137
  Black or African American | 0 | 1 | 1
  Hispanic or Latino | 3 | 0 | 3
  Asian | 4 | 8 | 12
Radiotherapy delivery modality [Number; unit: Participants]
  IMRT | 52 | 42 | 94
  3D-CRT | 35 | 21 | 56
  Missing | 2 | 1 | 3
Primary tumor site [Number; unit: Participants]
  Oropharynx/Larynx | 68 | 41 | 109
  Oral Cavity/Hypopharynx | 21 | 23 | 44
Nodal status [Number; unit: Participants] — N0: No regional lymph node metastasis. N+: Metastasis in one or more regional lymph nodes
  Participants
    N0 | 12 | 9 | 21
    N+ | 77 | 55 | 132
Tumor stage [Number; unit: Participants] — Staged according to the American Joint Committee on Cancer (AJCC) Staging Manual (6th edition).
  Participants
    T1-3 | 64 | 45 | 109
    T4 | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Local Regional Control Rate at 2 Years
Description: In this study participants were considered to be in local regional control (LRC) if there was no evidence of active disease in the previously affected/irradiated head-and-neck area. LRC could be achieved at any time following completion of treatment unless disease progression in the local-regional area occurred or the participant received subsequent anti-tumor therapy. Local regional control rate is defined as the Kaplan-Meier (KM) estimate of the proportion of participants with local regional control.
Time Frame: 2 years
Population: Efficacy Analysis Set (all randomized participants who received at least 1 dose of protocol-specified treatment according to treatment randomization regardless of treatment received.)
Measure: Number (95% Confidence Interval); unit: proportion of paticipants
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 63
proportion of paticipants | 0.61 [0.50 to 0.71] | 0.68 [0.54 to 0.78]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; Difference in Kaplan-Meier estimate = -0.07, 95% CI 2-sided [-0.23 to 0.09] — The difference between the treatment groups is calculated as panitumumab plus chemoradiation minus chemoradiotherapy alone

2. Secondary Outcome: Local Regional Control Rate at 6 Months and 12 Months
Description: Participants were considered to be in local regional control (LRC) if there was no evidence of active disease in the previously affected/irradiated head-and-neck area. LRC could be achieved at any time following completion of treatment unless disease progression in the local-regional area occurred or the participant received subsequent anti-tumor therapy. Local regional control rate is defined as the Kaplan-Meier (KM) estimate of the proportion of participants with local regional control.
Time Frame: 6 months and 12 months
Population: Efficacy Analysis Set
Measure: Number (95% Confidence Interval); unit: proportion of paticipants
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 63
proportion of paticipants
  6 months | 0.70 [0.59 to 0.79] | 0.73 [0.60 to 0.83]
  12 months | 0.66 [0.55 to 0.75] | 0.70 [0.56 to 0.80]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Difference between treatment groups at 6 months; Test type: Superiority or Other; Difference in Kaplan-Meier estimate = -0.03, 95% CI 2-sided [-0.18 to 0.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Difference between treatment groups at 12 months; Test type: Superiority or Other; Difference in Kaplan-Meier estimate = -0.03, 95% CI 2-sided [-1.09 to 0.12] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Duration of Local-regional Control
Description: Duration of local regional control is calculated from the first day of any study treatment (radiotherapy, chemotherapy, or panitumumab) administration to the date of first local-regional failure or to death due to any cause (whichever occurs first). Local-regional failure includes persistent disease and local-regional recurrence of disease. Participants who did not meet the criteria for LRC recurrence after achieving a response by the analysis data cutoff date were censored at their last evaluable disease assessment date. Participants who never achieved LRC were considered to have a duration of 0.
Time Frame: From first dose up to 37 months
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 63
months | 33.7 [28.8 to NA] — Upper limit could not be estimated due to the low number of events | NA [NA to NA] — Median could not be estimated due to the low number of events.
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; p = 0.3106, Regression, Cox; Hazard Ratio (HR) = 1.328, 95% CI 2-sided [0.767 to 2.299] — Hazard ratio is presented as panitumumab plus chemoradiation:chemoradiotherapy alone

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival time is defined as time from the first day of any study treatment to date of first progresive disease using a modified version of the World Health Organization (WHO) criteria or death.
  Progressive Disease is defined as at least a 25% increase in the size of index lesions or unequivocal progression of existing non-index lesions or the presence of one or more new lesions.
  Participants not meeting these criteria by the cutoff date were censored at their last evaluable disease assessment date.
Time Frame: From first dose date to 37 months
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 63
months | NA [24.3 to NA] — Could not be estimated due to the low number of events | NA [25.6 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; p = 0.6069, Regression, Cox; Hazard Ratio (HR) = 1.150, 95% CI 2-sided [0.675 to 1.961] — Hazard ratio is presented as panitumumab plus chemoradiation:chemoradiotherapy alone

5. Secondary Outcome: Overall Survival
Description: Survival time is defined as time from the first day of any study treatment to date of death. Participants who had not died by the cutoff date were censored at their last contact date.
Time Frame: From first dose date up to 37 months
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 63
months | 33.7 [32.2 to NA] — Could not be estimated due to the low number of events | NA [34.6 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; p = 0.1223, Regression, Cox; Hazard Ratio (HR) = 1.628, 95% CI 2-sided [0.877 to 3.019] — Hazard ratio is presented as panitumumab plus chemoradiation:chemoradiotherapy alone

6. Secondary Outcome: Percentage of Participants With an Objective Response at 6 Months
Description: Objective response by 6 months is defined as a complete response or partial response based on central review of scans using a a modification of the WHO criteria during the first 6 months.
  Complete Response (CR): Disappearance of all index and non-index lesions and no new lesions. Partial Response (PR): At least a 50% decrease in the size of index lesions with no progression in non-index lesions, or the disappearance of all index lesions and persistence of 1 or more non-index lesions not qualifying for either CR or progressive disease and no new lesions.
Time Frame: 6 months
Population: Evaluable for Central Tumor Response Analysis Set: the subset of participants in the Efficacy Analysis Set with at least one bi-dimensionally measurable lesion at baseline using a modified version of the WHO criteria per blinded central review.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 62
percentage of participants | 71.26 [60.57 to 80.46] | 82.26 [70.47 to 90.80]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; p = 0.1737, Regression, Logistic; Odds Ratio (OR) = 0.535, 95% CI 2-sided [0.217 to 1.262] — The odds ratio is defined as the odds of having an overall response in the panitumumab plus chemoradiation arm relative to the odds in the chemoradiotherapy alone arm
Statistical Analysis 2: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; Difference in rate = -10.99, 95% CI 2-sided [-24.56 to 4.14] — Difference is presented as the rate in panitumumab plus chemoradiation arm minus the rate in chemoradiotherapy alone arm

7. Secondary Outcome: Percentage of Participants With a Complete Response at 6 Months
Description: Response assessment based on central review of scans using a a modification of the WHO criteria, during the first 6 months. Complete Response is defined as the disappearance of all index and non-index lesions and no new lesions.
Time Frame: 6 months
Population: Evaluable for Central Tumor Response Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Plus Chemoradiation | Chemoradiotherapy Alone
Number analyzed (Participants) | 87 | 62
percentage of participants | 20.69 [12.75 to 30.71] | 19.35 [10.42 to 31.37]
Statistical Analysis 1: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; p = 1.0000, Regression, Logistic; Odds Ratio (OR) = 1.087, 95% CI 2-sided [0.448 to 2.712] — The odds ratio is defined as the odds of having a complete response in the panitumumab plus chemoradiation arm relative to the odds in the chemoradiotherapy alone arm
Statistical Analysis 2: Comparison: Panitumumab Plus Chemoradiation vs Chemoradiotherapy Alone; Test type: Superiority or Other; Difference in rate = 1.33, 95% CI 2-sided [-13.23 to 14.71] — [estimate comment as in outcome 6, analysis 2]

ADVERSE EVENTS:
Time Frame: The median reporting period was around 82 days in the Panitumumab Plus Chemoradiation arm, and around 80 days in the Chemoradiotherapy Alone arm.
Description: The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency in either treatment arm.
Arm/Group | Panitumumab Plus Chemoradiation | Chemotherapy Plus Radiotherapy
Serious Adverse Events (participants affected / at risk) | 37/87 | 20/63
Other Adverse Events (participants affected / at risk) | 87/87 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemoradiation (N=87) | Chemotherapy Plus Radiotherapy (N=63)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 6 | 4
Glossitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 3 | 1
Mucosal inflammation (General disorders) | 6 | 1
Pyrexia (General disorders) | 5 | 1
Bacteraemia (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 5 | 0
Stomatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 3
Renal failure acute (Renal and urinary disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Chemoradiation (N=87) | Chemotherapy Plus Radiotherapy (N=63)
Anaemia (Blood and lymphatic system disorders) | 21 | 13
Neutropenia (Blood and lymphatic system disorders) | 6 | 8
Deafness (Ear and labyrinth disorders) | 4 | 7
Tinnitus (Ear and labyrinth disorders) | 8 | 12
Constipation (Gastrointestinal disorders) | 34 | 21
Diarrhoea (Gastrointestinal disorders) | 18 | 7
Dry mouth (Gastrointestinal disorders) | 41 | 33
Dyspepsia (Gastrointestinal disorders) | 12 | 6
Dysphagia (Gastrointestinal disorders) | 55 | 40
Nausea (Gastrointestinal disorders) | 45 | 36
Odynophagia (Gastrointestinal disorders) | 21 | 19
Oral pain (Gastrointestinal disorders) | 9 | 3
Stomatitis (Gastrointestinal disorders) | 15 | 11
Vomiting (Gastrointestinal disorders) | 29 | 21
Asthenia (General disorders) | 12 | 7
Fatigue (General disorders) | 19 | 18
Mucosal inflammation (General disorders) | 71 | 45
Oedema peripheral (General disorders) | 5 | 2
Pain (General disorders) | 8 | 1
Pyrexia (General disorders) | 10 | 7
Candidiasis (Infections and infestations) | 11 | 1
Device related infection (Infections and infestations) | 5 | 0
Infection (Infections and infestations) | 9 | 0
Oral candidiasis (Infections and infestations) | 10 | 7
Radiation skin injury (Injury, poisoning and procedural complications) | 58 | 52
Blood creatinine increased (Investigations) | 6 | 5
Haemoglobin decreased (Investigations) | 0 | 5
Weight decreased (Investigations) | 37 | 28
Decreased appetite (Metabolism and nutrition disorders) | 20 | 19
Dehydration (Metabolism and nutrition disorders) | 6 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Dizziness (Nervous system disorders) | 5 | 7
Dysgeusia (Nervous system disorders) | 21 | 27
Headache (Nervous system disorders) | 5 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 5 | 3
Depression (Psychiatric disorders) | 6 | 0
Insomnia (Psychiatric disorders) | 13 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Acne (Skin and subcutaneous tissue disorders) | 16 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 10 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 13 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 1
Erythema (Skin and subcutaneous tissue disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 0
Rash (Skin and subcutaneous tissue disorders) | 40 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 5 | 0
Hypotension (Vascular disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.